CLINICAL TRIAL: NCT04107675
Title: A Phase IIa Multi-Center, Randomized, Single-Blind Safety Study of Liposomal Cyclosporine A to Treat Bronchiolitis Obliterans Syndrome Following Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: A Safety Study of Liposomal Cyclosporine A to Treat Bronchiolitis After Hematopoietic Transplant (BOSTON-4)
Acronym: BOSTON-4
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to the low number of patients recruited and the slow enrollment pace of patients, on 18 March 2022, the sponsor decided to terminate the BOSTON-4 safety and tolerability trial ahead of time.
Sponsor: Zambon SpA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BT - L-CsA - 201 - SCT; 2019-000718-13 (EudraCT Number)
Record Dates: First submitted 2019-09-25; First posted 2019-09-27 (Actual); Results first posted 2023-10-03 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-09

CONDITIONS: Bronchiolitis Obliterans Syndrome (BOS); GVHD, Chronic; Stem Cell Transplant Complications
Keywords: stem cell; hematopoietic transplant
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Who Masked: Participant
Masking Description: This was a single-blind trial. Due to the different appearance of the 3 tested strengths of IMP, a full blinding of the study was not possible. Only the randomized study patients were blinded to study treatment assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- L-CsA 10 mg plus Standard of Care (Experimental): Liposomal Cyclosporine A 10 mg (10 mg/2.5 mL) bid, once in the morning and once in the evening, for up to 12 weeks.
  The inhalations were scheduled to be taken approximately 12 hours (but not less than 6 hours) apart, eg, at 08:00 and 20:00 each day. Nebulization time per inhalation dose was approximately 8 to 13 minutes for the 0- and 10-mg doses.
  Standard of care included prophylaxis against common opportunistic infections, immunosuppression, and any other chronic medication
  Interventions: Drug: Liposomal Cyclosporine A
- L-CsA 5 mg plus Standard of Care (Experimental): Liposomal Cyclosporine A 5 mg (5 mg/1.25 mL) bid, once in the morning and once in the evening, for up to 12 weeks. The inhalations were scheduled to be taken approximately 12 hours (but not less than 6 hours) apart, eg, at 08:00 and 20:00 each day. Nebulization time per inhalation dose was approximately 5 to 10 minutes for the 5-mg dose.
  Standard of care included prophylaxis against common opportunistic infections, immunosuppression, and any other chronic medication
  Interventions: Drug: Liposomal Cyclosporine A
- Liposomal Placebo plus Standard of Care (Placebo Comparator): Liposomal Placebo 2.5 mL (0 mg L-CsA/2.5 mL) bid, once in the morning and once in the evening, for up to 12 weeks.
  The inhalations were scheduled to be taken approximately 12 hours (but not less than 6 hours) apart, eg, at 08:00 and 20:00 each day. Nebulization time per inhalation dose was approximately 8 to 13 minutes for the 0- and 10-mg doses. Standard of care included prophylaxis against common opportunistic infections, immunosuppression, and any other chronic medication
  Interventions: Drug: Liposomal Placebo

INTERVENTIONS:
Drug: Liposomal Cyclosporine A — Liposomal Cyclosporine A is administered at different dosages in the first two arms (10 mg bid and 5 mg bid, respectively) with a new technology of nebulizing liquid drugs, creating an aerosol with a low ballistic momentum and a high percentage of droplets in a respirable size range of 3-5 μm
  Other Names: L-CsA
  Arms: L-CsA 10 mg plus Standard of Care; L-CsA 5 mg plus Standard of Care
Drug: Liposomal Placebo — Liposomal Placebo is administered with the same new technology of nebulizing liquid drugs used for L-CsA, creating an aerosol with a low ballistic momentum and a high percentage of droplets in a respirable size range of 3-5 μm
  Other Names: Placebo
  Arms: Liposomal Placebo plus Standard of Care

SUMMARY:
Primary Objective:

The primary objective of this study is to assess the tolerability and safety of two dose levels of aerosolized L-CsA vs placebo in addition to SoC therapy for BOS in adult allo-HSCT recipients.

Secondary Objectives:

The secondary objectives of this study are to assess PK and exploratory efficacy and quality of life of two dose levels of aerosolized L-CsA vs placebo in addition to SoC therapy for BOS in adult allo-HSCT recipients.

DETAILED DESCRIPTION:
This is a Phase II prospective, multi-center, single-blind, randomized clinical trial evaluating safety and tolerability in adult recipients of an allo-HSCT with BOS. Twenty-four patients were planned for enrollment; but, at the time of the premature termination of this study, a total of 11 patients were screened for the study, of whom 5 patients did not fulfill the inclusion criteria and 6 patients were randomly allocated 1:1:1 in 3 treatment groups (L-CsA 10 mg + SoC, L-CsA 5 mg + SoC, or placebo + SoC).

A total of 18 centers in 3 countries (France, Germany, and Spain) in Europe were initiated for this multi-center study.

IMP was administered for up to 12 weeks treatment period. With low patient recruitment, the BOSTON-4 safety and tolerability study was terminated early by the sponsor on 18 March 2022. This decision was made after a careful and due diligent analysis performed by Zambon of the study status and considering the impact of coronavirus disease 2019 (COVID-19) pandemic on sites activities. From the beginning of the study, in December 2019, only 6 patients were randomized. So it was estimated that continuing the trial with the current protocol and setting would have taken another 9 years for the study to complete.

ELIGIBILITY:
Inclusion Criteria:

1. Age >/= 18 years
2. Patient must have a history of allogeneic HSCT, regardless of source of stem cell or donor or indication for allogeneic HSCT
3. Documented diagnosis of chronic Graft versus Host Disease (cGvHD) in any organ other than the lung. If BOS is the only manifestation of cGvHD, lung biopsy must have been performed before entering the trial to confirm BOS diagnosis.
4. Confirmed diagnosis of BOS Score 1 [Jagasia et al. 2015] within > 6 months and < 3 years after allo-HSCT:

   FEV1/FVC < 0.7 at Screening Visit AND Post-bronchodilator FEV1 >/= 60 and ≤ 79% predicted at Screening Visit AND
   * 10% decline of FEV1 % predicted within 24 months prior to Screening Visit AND Absence of acute infection in the respiratory tract.
5. Patient must be capable of understanding the purposes and risks of the study, has given written informed consent, and agrees to comply with the study requirements.
6. Patient is capable of aerosol inhalation.
7. Women of childbearing potential must have a negative serum or urine pregnancy test at screening and at randomization visit.

Exclusion Criteria:

1. Active bacterial, viral (as confirmed by multiplex PCR) or fungal infection not successfully resolved at least 4 weeks prior to the Screening Visit.
2. Chronic renal dysfunction with serum creatinine >/= 2.5 mg/dL or need for renal dialysis.
3. Chronic hepatic dysfunction with serum total bilirubin > 5x upper limit of normal (ULN), transaminases > 5x ULN, or alkaline phosphatase > 5x ULN.
4. Evidence of relapse of the primary malignancy which warranted allogeneic bone marrow transplant.
5. Use of azithromycin within 4 weeks prior to Randomization (Visit 1).
6. Use of zafirlukast during the study period.
7. Chronic oxygen use or use of non-invasive ventilation.
8. Active smokers (i.e. any kind of inhaled nicotine consumption).
9. Pregnant women or women who are unwilling to use appropriate birth control to avoid pregnancy over the course of the clinical trial.
10. Women who are currently breastfeeding.
11. Known hypersensitivity to L-CsA or to cyclosporine A.
12. Patients who do not tolerate administration of inhaled bronchodilators (e.g., salbutamol).
13. Patients with life-expectancy of less than 6 months.
14. Treatments with other Investigational Medicinal Products (IMPs) or previous therapies within four weeks or five times half-life of the drug, whichever is longer prior to screening and during the study. Participation in registries, considering the before, is allowed.
15. Psychiatric disorders or altered mental status precluding understanding of the informed consent process and/or completion of the necessary procedures.
16. Any co-existing medical condition that in the Investigator's judgment will substantially increase the risk associated with the patient's participation in the clinical trial.
17. Pre-scheduled hospitalizations, surgeries or interventions planned to be performed after obtaining Informed Consent for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2020-02-11 (Actual); Primary Completion 2022-06-16 (Actual); Study Completion 2022-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paola Castellani, MD, Study Director — Zambon SpA, Chief Medical Officer
Locations (17):
- France (8):
  - CHU Hôpital Sud, Amiens
  - Centre Hospitalier Universitaire d'Angers, Angers
  - Centre Hospitalier Universitaire Grenoble Alpes - Hopital Albert Michallon, La Tronche
  - Centre Hospitalier Régional Universitaire de Lille (CHRU) - Hôpital Claude Huriez, Lille
  - CHU de Nancy, Hopital Brabois, Nancy
  - CHU de Nantes - Hotel-Dieu, Nantes
  - Hopital Saint Louis, Paris
  - CHU Hopitaux de Bordeaux - Hôpital Haut-Lévêque, Pessac
- Germany (4):
  - Universitätsklinikum Köln, Cologne
  - St.-Johannes-Hospital, Dortmund
  - Universitätsklinikum Carl Gustav Carus, Dresden
  - Universitätsklinikum Münster, Münster
- Spain (5):
  - Hospital Clinic i Provincial, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Clinico Universitario de Valencia, Valencia
  - Hospital Universitari i Politècnic La Fe, Valencia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From the start of the trial, only 6 patients were randomized. With low patient recruitment, the BOSTON-4 safety and tolerability study was terminated early on 18 March 2022. This decision was made after a careful and due diligent analysis performed by Zambon of the study status and considering the impact of coronavirus disease 2019 (COVID-19) pandemic on sites activities. So, due to this low recruitment, the Sponsor decided to early terminate the trial, on 18 March 2022.
Groups:
- L-CsA 10 mg Plus Standard of Care: Liposomal Cyclosporine A 10 mg (10 mg/2.5 mL) bid, once in the morning and once in the evening, for up to 12 weeks.
  The inhalations were scheduled to be taken approximately 12 hours (but not less than 6 hours) apart, eg, at 08:00 and 20:00 each day. Nebulization time per inhalation dose was approximately 8 to 13 minutes for the 0- and 10-mg doses.
  Standard of care included prophylaxis against common opportunistic infections, immunosuppression, and any other chronic medication
  Liposomal Cyclosporine A: Liposomal Cyclosporine A is administered at different dosages in the first two arms (10 mg bid and 5 mg bid, respectively) with a new technology of nebulizing liquid drugs, creating an aerosol with a low ballistic momentum and a high percentage of droplets in a respirable size range of 3-5 μm
- L-CsA 5 mg Plus Standard of Care: Liposomal Cyclosporine A 5 mg (5 mg/1.25 mL) bid, once in the morning and once in the evening, for up to 12 weeks. The inhalations were scheduled to be taken approximately 12 hours (but not less than 6 hours) apart, eg, at 08:00 and 20:00 each day. Nebulization time per inhalation dose was approximately 5 to 10 minutes for the 5-mg dose.
  Standard of care included prophylaxis against common opportunistic infections, immunosuppression, and any other chronic medication
  Liposomal Cyclosporine A: Liposomal Cyclosporine A is administered at different dosages in the first two arms (10 mg bid and 5 mg bid, respectively) with a new technology of nebulizing liquid drugs, creating an aerosol with a low ballistic momentum and a high percentage of droplets in a respirable size range of 3-5 μm
- Liposomal Placebo Plus Standard of Care: Liposomal Placebo 2.5 mL (0 mg L-CsA/2.5 mL) bid, once in the morning and once in the evening, for up to 12 weeks.
  The inhalations were scheduled to be taken approximately 12 hours (but not less than 6 hours) apart, eg, at 08:00 and 20:00 each day. Nebulization time per inhalation dose was approximately 8 to 13 minutes for the 0- and 10-mg doses. Standard of care included prophylaxis against common opportunistic infections, immunosuppression, and any other chronic medication
  Liposomal Placebo: Liposomal Placebo is administered with the same new technology of nebulizing liquid drugs used for L-CsA, creating an aerosol with a low ballistic momentum and a high percentage of droplets in a respirable size range of 3-5 μm
Period: Overall Study
Arm/Group | L-CsA 10 mg Plus Standard of Care | L-CsA 5 mg Plus Standard of Care | Liposomal Placebo Plus Standard of Care
Started | 2 | 2 | 2
Completed | 2 | 2 | 2
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set (SAF) was defined as all randomized patients who had received a partial dose of IMP at least once.
Groups:
- Total: Total of all reporting groups
Arm/Group | L-CsA 10 mg Plus Standard of Care | L-CsA 5 mg Plus Standard of Care | Liposomal Placebo Plus Standard of Care | Total
Number analyzed (Participants) | 2 | 2 | 2 | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 2 | 6
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.5 (0.71) | 63.0 (0.00) | 46.0 (12.73) | 54.8 (9.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 1 | 3
  Male | 2 | 0 | 1 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1 | 2
  Not Hispanic or Latino | 0 | 0 | 1 | 1
  Unknown or Not Reported | 2 | 1 | 0 | 3
Region of Enrollment [Number; unit: participants]
  France | 1 | 1 | 0 | 2
  Germany | 1 | 0 | 1 | 2
  Spain | 0 | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Local Tolerability Events of Interest From Baseline to Visit 3 (Week 4)
Description: The local tolerability events of interest taken into consideration were: Cough, Wheezing, Bronchospasm, Throat irritation and Change from baseline in FEV1 to Visit 3.
Time Frame: at Week 4 (visit 3)
Population: as for baseline characteristics
Measure: Number; unit: number of local events
Arm/Group | L-CsA 10 mg Plus Standard of Care | L-CsA 5 mg Plus Standard of Care | Liposomal Placebo Plus Standard of Care
Number analyzed (Participants) | 2 | 2 | 2
number of local events
  Any Local Tolerability Event | 1 | 5 | 4
  Cough | 0 | 1 | 1
  Wheezing | 0 | 0 | 0
  Bronchospasm | 0 | 0 | 0
  Throat irritation | 1 | 3 | 2
  Change in FEV1 | 0 | 1 | 1

2. Primary Outcome: Number of Participants With AE and sAE of Different Level of Severity During the First 4 Weeks of Treatment
Description: An adverse event (AE) is any untoward medical occurrence after exposure to a medicine, which is not necessarily caused by that medicine. An adverse event can therefore be any unfavourable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.
  A serious adverse event is an adverse event that results in death, is life-threatening, requires hospitalisation or prolongation of existing hospitalisation, results in persistent or significant disability or incapacity, or is a birth defect.
Time Frame: During the first 4 weeks of treatment
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | L-CsA 10 mg Plus Standard of Care | L-CsA 5 mg Plus Standard of Care | Liposomal Placebo Plus Standard of Care
Number analyzed (Participants) | 2 | 2 | 2
Participants
  Any TEAEs | 1 | 1 | 1
  Mild TEAEs | 1 | 1 | 1
  Moderate TEAEs | 0 | 0 | 0
  Severe TEAEs | 0 | 0 | 0
  Serious TEAEs | 0 | 0 | 0
  Related TEAEs | 1 | 1 | 1
  COVID-19 related TEAEs | 0 | 0 | 0
  Patients discontinued study due to TEAEs | 0 | 0 | 0
  Patients discontinued treatment due to TEAEs | 0 | 0 | 0
  TEAEs Leading to Death | 0 | 0 | 0

3. Secondary Outcome: Number of Local Tolerability Events of Interest From Baseline to Week 12
Description: as for outcome 1
Time Frame: at Week 12
Population: as for baseline characteristics
Measure: Number; unit: number of events
Arm/Group | L-CsA 10 mg Plus Standard of Care | L-CsA 5 mg Plus Standard of Care | Liposomal Placebo Plus Standard of Care
Number analyzed (Participants) | 2 | 2 | 2
number of events
  Any Local Tolerability Event | 1 | 7 | 6
  Cough | 0 | 2 | 2
  Wheezing | 0 | 0 | 0
  Bronchospasm | 0 | 0 | 0
  Throat irritation | 1 | 4 | 3
  Change in FEV1 | 0 | 1 | 1

4. Secondary Outcome: Number of Participants With AE and sAE of Different Level of Severity During the First 12 Weeks of Treatment
Description: as for outcome 2
Time Frame: During the first 12 weeks of treatment
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | L-CsA 10 mg Plus Standard of Care | L-CsA 5 mg Plus Standard of Care | Liposomal Placebo Plus Standard of Care
Number analyzed (Participants) | 2 | 2 | 2
Participants
  Any TEAEs | 2 | 1 | 1
  Mild TEAEs | 2 | 1 | 1
  Moderate TEAEs | 1 | 0 | 0
  Severe TEAEs | 0 | 0 | 0
  Serious TEAEs | 1 | 0 | 0
  Related TEAEs | 1 | 1 | 1
  COVID-19 related TEAEs | 0 | 0 | 0
  Patients discontinued study due to TEAEs | 0 | 0 | 0
  Patients discontinued treatment due to TEAEs | 1 | 0 | 0
  TEAEs Leading to Death | 0 | 0 | 0

5. Secondary Outcome: CsA Whole Blood Concentrations and CsA Whole Blood Trough Levels
Description: Whole Blood concentrations (Week 0) are at pre-dose, directly after end of inhalation, 15, 30, and 45 minutes, and 1, 1.5, 2, and 4 hours after end of inhalation, and whole blood trough levels (CsA concentration) at Weeks 2, 4, 8, and 12 were calculated.
Time Frame: Weeks 0 (pre-dose, directly after end of inhalation, 15, 30, 45, 60 min, 1.5 h, 2h, 4h), 2, 4, 8, and 12
Population: The Full Analysis Set (FAS) was defined as all randomized patients for whom at least
  1 post-baseline measurement of an efficacy outcome measure (ie, spirometry or quality of life measures) was available. For spirometry measures, baseline corresponded to the assessment at randomization visit (Visit 1) prior to inhalation of IMP.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | L-CsA 10 mg Plus Standard of Care | L-CsA 5 mg Plus Standard of Care | Liposomal Placebo Plus Standard of Care
Number analyzed (Participants) | 2 | 2 | 2
ng/ml
  Week 0 - predose | 12.2115 (17.26967) | 0.0000 (0.0000) | 11.7750 (16.65236)
  Directly after end of inhalation | 84.6510 (69.82821) | 19.3420 (15.91980) | 12.1760 (17.21946)
  15 min | 73.5110 (59.82123) | 30.0500 (24.34003) | 11.2440 (15.90142)
  30 min | 68.3640 (60.56228) | 26.9400 (22.19184) | 13.1780 (18.63651)
  45 min | 70.1555 (64.88483) | 23.2780 (18.52761) | 13.3145 (18.82955)
  1 hour: number analyzed (Participants) | 1 | 2 | 2
  1 hour | 117.8030 (NA) — Standard Deviation is not calculable for 1 participant | 19.4395 (18.15638) | 14.0835 (19.91708)
  1.5 hours: number analyzed (Participants) | 1 | 2 | 2
  1.5 hours | 115.4350 (NA) — Standard Deviation is not calculable for 1 participant | 16.0300 (13.34876) | 13.0425 (18.44488)
  2 hours | 67.0700 (71.46587) | 13.4045 (10.80530) | 10.9615 (15.50190)
  4 hours | 33.3425 (35.73506) | 8.3950 (8.09920) | 7.6615 (10.83500)
  Whole Blood Trough Levels - Week 2 | 48.6725 (64.65148) | 4.6365 (3.62534) | 6.0500 (8.55599)
  Whole Blood Trough Levels - Week 4 | 16.2465 (17.33048) | 16.8475 (21.28745) | 6.3000 (8.90955)
  Whole Blood Trough Levels - Week 8 | 18.7280 (26.48539) | 9.0405 (3.16855) | 4.9500 (7.00036)
  Whole Blood Trough Levels - Week 12: number analyzed (Participants) | 2 | 1 | 2
  Whole Blood Trough Levels - Week 12 | 23.0195 (32.55449) | 0.0000 (NA) — Standard Deviation is not calculable for 1 participant | 4.9500 (7.00036)

ADVERSE EVENTS:
Time Frame: Throughout the complete clinical trial period, i.e. up to week 14 (visit 6 / EoS).
Description: Please note that if a patient has multiple occurrences of an AE, the patient is presented only once in the respective patient count
Arm/Group | L-CsA 10 mg Plus Standard of Care | L-CsA 5 mg Plus Standard of Care | Liposomal Placebo Plus Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 1/2 | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 2/2 | 1/2 | 1/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | L-CsA 10 mg Plus Standard of Care (N=2) | L-CsA 5 mg Plus Standard of Care (N=2) | Liposomal Placebo Plus Standard of Care (N=2)
moderate acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | L-CsA 10 mg Plus Standard of Care (N=2) | L-CsA 5 mg Plus Standard of Care (N=2) | Liposomal Placebo Plus Standard of Care (N=2)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
From the beginning of the trial, only 6 patients were enrolled. Due to the low number of patients recruited so far and the slow enrolment pace of patients, on 18 March 2022, the sponsor decided to terminate the BOSTON-4 safety and tolerability trial early. This decision was made after the Sponsor performed a careful and due diligent analysis of the current study status and considered the impact of the coronavirus disease 2019 (COVID-19) pandemic on-site activities.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-04-30): https://cdn.clinicaltrials.gov/large-docs/75/NCT04107675/Prot_000.pdf
  • Statistical Analysis Plan (2022-02-25): https://cdn.clinicaltrials.gov/large-docs/75/NCT04107675/SAP_001.pdf